CLINICAL TRIAL: NCT02773693
Title: Treatment of Comorbid Sleep Disorders and Post Traumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of North Texas, Denton, TX (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); South Texas Veterans Health Care System (U.S. Federal Agency); Duke University (Other); Durham VA Medical Center (U.S. Federal Agency); Boston VA Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-13-2-0065; 1 I01 CX001136-01 (Other Grant/Funding Number: Veterans Affairs)
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Trauma; Insomnia; Nightmares
MeSH Terms: conditions — Wounds and Injuries; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CPT (Active Comparator): Cognitive Processing Therapy-cognitive only version (typically labeled CPT-C, but labeled CPT in this grant for simplicity) is a type of Cognitive Therapy addressing daytime symptoms of PTSD. This arm will have 12 twice-weekly sessions, followed by 6 weekly sessions.
  Interventions: Behavioral: Cognitive Processing Therapy-Cognitive Only (CPT); Behavioral: Continuation Cognitive Processing Therapy-Cognitive Only (CPT)
- CBTin+CPT (Active Comparator): Cognitive Behavioral Therapy of Insomnia and nightmares (CBTin) will be used to address nighttime symptoms of PTSD during 6 weekly sessions, followed by 12 twice-weekly sessions of CPT.
  Interventions: Behavioral: Cognitive Processing Therapy-Cognitive Only (CPT); Behavioral: Cognitive Behavioral Therapy of Insomnia and Nightmares (CBTin)
- CPT+CBTin (Active Comparator): 12 twice-weekly sessions of CPT followed by 6 sessions of CBTin.
  Interventions: Behavioral: Cognitive Processing Therapy-Cognitive Only (CPT); Behavioral: Cognitive Behavioral Therapy of Insomnia and Nightmares (CBTin)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy-Cognitive Only (CPT) — Twice weekly CPT over 6 weeks.
Behavioral: Cognitive Behavioral Therapy of Insomnia and Nightmares (CBTin) — Cognitive behavioral therapy of insomnia and nightmares weekly over 6 weeks.
  Arms: CBTin+CPT; CPT+CBTin
Behavioral: Continuation Cognitive Processing Therapy-Cognitive Only (CPT) — Once weekly continuation CPT over 6 weeks.
  Arms: CPT

SUMMARY:
The primary objective of the current study is to determine if providing cognitive-behavioral therapy of Insomnia and nightmares (CBTin) and Cognitive Processing Therapy of PTSD (CPT) results in greater PTSD and sleep symptom reduction than CPT only. A secondary objective is to determine if the sequencing of CBTl&N before or after CPT results in differential effects on PTSD and sleep symptom reduction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50.
* Chronic Insomnia, as defined by the Diagnostic and Statistical Manual-fifth edition (DSM-5) (American Psychiatric Association, 2013) assessed with Structured Clinical Interview for DSM-5 Sleep Disorders (SCISD).
* Chronic Nightmare Disorder, as defined by DSM-5, assessed with the SCISD.
* PTSD, as defined by DSM-5, assessed by Clinician-Administered Posttraumatic Stress Scale-5 (CAPS-5).
* Active duty military and recently discharged Veterans at Fort Hood eligible for treatment at Carl R. Darnall Army Medical Center (CRDAMC).
* History of having deployed in support of combat operations following 9/11, assessed by self-report.
* Stable on psychotropic and/or hypnotic medications and/or interventions for sleep (e.g., Continuous Positive Air Pressure for sleep apnea) administered by other providers for at least one month assessed by self-report and review of medical record.
* Willing to refrain from new behavioral health or medication treatment for issues pertaining to sleep, PTSD, or nightmares during participation in the study.
* Indication that the individual plans to be in the area for the 5 months following the first assessment.

Exclusion Criteria:

* Individuals who have been re-deployed from a theater of operation less than 3 months.
* Current suicide or homicide risk meriting crisis intervention as assessed by the Patient Health Questionnaire (PHQ-9), The Depressive Symptom Index - Suicidality Subscale (DSI-SS), or the Self-Injurious Thoughts and Behaviors Interview (SITBI).
* Inability to speak and read English.
* Moderate to severe brain damage, assessed by the inability to comprehend the baseline questionnaires.
* Pregnancy, assessed by self-report and review of medical record, because sleep disturbances due to pregnancy may be the result of different mechanisms and the proposed instruments and treatments have not been validated in this population.
* Current circadian rhythm, environmental, sleep deprivation, or hypersomnia sleep disorder, assessed by self-report because CBTin has not been validated in these populations.
* Other untreated sleep disorders to include individuals with clinically significant obstructive sleep apnea (Respiratory Disturbance Index >5/hr), periodic limb movement disorder (PLMD; >15/hr with arousals), nocturnal seizures, or a parasomnia (e.g., sleepwalking, confusional arousals, nocturnal eating and drinking syndrome), based on criteria from the International Classification of Sleep Disorders-third edition (American Academy of Sleep Medicine, 2013). Individuals meeting criteria for one of the above sleep disorders will be seen for clinical care at the CRDAMC Sleep Center. Once the aforementioned sleep disorder is stably treated, individuals meeting the study criteria for insomnia, nightmares, and PTSD can be reassessed for participation in this study.
* Sleep efficiency >85%, as assessed by the sleep diary.
* Serious mental health diagnosis (e.g., bipolar disorder or psychosis) assessed with review of baseline questionnaires, review of medical record, and/or Mini International Neuropsychiatric Interview (MINI 7.0 Mania module).
* Currently engaged in evidence-based psychotherapy for PTSD (i.e., Prolonged Exposure Therapy or Cognitive Processing Therapy) or Insomnia or nightmares (i.e., Cognitive Behavioral Therapy) by self-report and review of medical record.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2016-08; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS-5) | Change from baseline to 1-month post-treatment (i.e., after the completion of all 18 sessions, not to exceed 22 weeks from baseline).
  The CAPS-5 (Weathers, Litz, et al., 2013) is a structured diagnostic interview and gold standard for assessing PTSD. The scale also assesses social and occupational functioning, dissociation, and the validity of symptom reports. The CAPS was revised to match DSM-5. The CAPS was revised to accommodate the changes made in DSM-5, to reduce administration time, and to facilitate learning administration and scoring procedures. The CAPS-5 will be the primary outcome of PTSD symptom severity.

SECONDARY OUTCOMES:
PTSD Checklist -DSM-5 (PCL-5) | Change from baseline to 1-month post-treatment (i.e., after the completion of all 18 sessions, not to exceed 22 weeks from baseline).
  The PCL-5 (Weathers, Blake, et al., 2013) is a 20-item self-report measure designed to assess PSTSD symptoms as defined by the DSM-5. The PCL-5 will be the secondary outcome of PTSD symptom severity.
Sleep Diary Sleep Efficiency | Change from baseline to 1-month post-treatment (i.e., after the completion of all 18 sessions, not to exceed 22 weeks from baseline).
  Sleep diaries will be used for seven days to measure subjective sleep patterns (Carney et al., 2012). Participants will be asked to make daily diary entries with an estimate of their sleep the night before (e.g., bedtime, sleep onset). Questions will also assess nightmare frequency and severity. Average sleep efficiency ((total sleep time/time in bed) x 100) derived from the sleep diaries will be the primary outcome of insomnia symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Taylor, Ph.D., Principal Investigator — University of North Texas Health Science Center
Locations (1):
- Carl R. Darnall Army Medical Center, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor DJ, Pruiksma KE, Mintz J, Slavish DC, Wardle-Pinkston S, Dietch JR, Dondanville KA, Young-McCaughan S, Nicholson KL, Litz BT, Keane TM, Peterson AL, Resick PA; Consortium to Alleviate PTSD. Treatment of comorbid sleep disorders and posttraumatic stress disorder in U.S. active duty military personnel: A pilot randomized clinical trial. J Trauma Stress. 2023 Aug;36(4):712-726. doi: 10.1002/jts.22939. Epub 2023 Jun 15. PMID 37322836
- [Derived] Miles SR, Pruiksma KE, Slavish D, Dietch JR, Wardle-Pinkston S, Litz BT, Rodgers M, Nicholson KL, Young-McCaughan S, Dondanville KA, Nakase-Richardson R, Mintz J, Keane TM, Peterson AL, Resick PA, Taylor DJ; Consortium to Alleviate PTSD. Sleep disorder symptoms are associated with greater posttraumatic stress and anger symptoms in US Army service members seeking treatment for posttraumatic stress disorder. J Clin Sleep Med. 2022 Jun 1;18(6):1617-1627. doi: 10.5664/jcsm.9926. PMID 35197191